CLINICAL TRIAL: NCT03381352
Title: Phase II Study of IMRT Radiotherapy Concurrent Chemothrerapy for Anal Cancer
Brief Title: Study of IMRT Radiotherapy Concurrent Chemothrerapy for Anal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LI Ning, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-MX2015-014
Record Dates: First submitted 2017-12-13; First posted 2017-12-22 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Anal Cancer
Keywords: Radiotherapy; Anal cancer; IMRT
MeSH Terms: conditions — Anus Neoplasms | interventions — Capecitabine; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemo-radiotherapy with IMRT technique (Experimental): Radiotherapy with IMRT technique concurrent with Capecitabine and MMC chemotherapy
  Interventions: Radiation: Chemo-radiotherapy with IMRT technique; Drug: Capecitabine; Drug: Mitomycin C

INTERVENTIONS:
Radiation: Chemo-radiotherapy with IMRT technique — IMRT radiation technique; 50.4-54Gy/25F
Drug: Capecitabine — Capecitabine 825mg/m2 PO BID
Drug: Mitomycin C — Mitomycin C 10mg/m2 D1,29 iv

SUMMARY:
The purpose of this study is to evaluate the efficacy and adverse events of intensity modulated radiation therapy (IMRT) concurrent with chemotherapy for anal squamous carcinoma. All enrolled anal squamous carcinoma patients are intented to receive IMRT concurrent with Capecitabine + mitomycin ± cetuximab targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* CT/MRI diagnosed stage cT1-4N0-3;
* Histologically confirmed anal squamous carcinoma;
* KPS >= 70
* Adequate organ function;
* No previous radiotherapy or chemotherapy;
* No surgery.

Exclusion Criteria:

* Previous malignant cancer history;
* Allegic to 5-fu or MMC

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | 8 weeks after IMRT
  To evaluate response rate of IMRT with chemotherapy

SECONDARY OUTCOMES:
Adverse events | from start of IMRT to 8 weeks after IMRT
  To assess the adverse events of IMRT with chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese academy of medical sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No